CLINICAL TRIAL: NCT00862563
Title: A Double-Blind, Placebo-Controlled, Parallel Group Design Trial of; Levetiracetam, Zonisamide, Topiramate, and Placebo Control for the Treatment of Alcohol Dependent Subjects.
Brief Title: Interdisciplinary Study of Two Novel Anticonvulsants in Alcoholism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment goals could not be met before ending of funding for this project.
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Dominic Ciraulo, Department Chair, Psychiatry, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAA-CIR-AA015923; P60AA013759 (NIH); 1R01AA015923 (NIH)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Alcoholism; Alcohol Dependence; Alcohol Abuse
Keywords: Alcoholism; Alcohol Dependence; Alcohol Abuse; Substance Abuse; Alcoholic Intoxication
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Alcoholic Intoxication | interventions — Topiramate; Zonisamide; Levetiracetam; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Zonisamide (Experimental): Encapsulated zonisamide with a target maintenance doses of 400 mg/day administered as 4 capsules per day.
  Interventions: Drug: Zonisamide
- Levetiracetam (Experimental): Encapsulated levetiracetam with a target maintenance doses of 2000 mg/day administered as 4 capsules per day .
  Interventions: Drug: Levetiracetam
- Topiramate (Active Comparator): Encapsulated topiramate with a target maintenance doses of 300 mg/day administered as 4 capsules per day .
  Interventions: Drug: Topiramate
- Sugar Pill (Placebo Comparator): Encapsulated sugar pill with a target maintenance dose administered as 4 capsules per day.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Topiramate — Topiramate will be administered orally twice daily beginning on Day 1, Week 1 and continue through Day 7, Week 14. Subjects will be dose titrated as tolerated to a target doses 300 mg topiramate.
  Other Names: Topamax
  Arms: Topiramate
Drug: Zonisamide — Zonisamide will be administered orally twice daily beginning on Day 1, Week 1 and continue through Day 7, Week 14. Subjects will be dose titrated as tolerated to a target doses of 2000 400 mg of zonisamide.
  Other Names: zonegran
  Arms: Zonisamide
Drug: Levetiracetam — Levetiracetam will be administered orally twice daily beginning on Day 1, Week 1 and continue through Day 7, Week 14. Subjects will be dose titrated as tolerated to a target doses of 2000 mg levetiracetam capsules.
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Sugar Pill — Matched placebo will be administered orally twice daily beginning on Day 1, Week 1 and continue through Day 7, Week 14.
  Other Names: Placebo
  Arms: Sugar Pill

SUMMARY:
This is a double-blind, placebo-controlled, parallel group design study with 4 treatment groups; levetiracetam, zonisamide, topiramate, and placebo control. Subjects will receive study medications for 14 weeks. Potential subjects will be initially screened for interest in study participation and alcohol consumption level to determine basic eligibility by telephone, or in person. Individuals who meet telephone screening criteria will be scheduled for a clinic appointment to obtain informed consent and conduct screening assessments. Subjects who report average drinks per day that are within the guidelines for safe levels of alcohol consumption (i.e. 2 drinks/ day males; 1 drink/day females-HHS standard) in the two weeks prior to screening will be excluded. Subjects meeting screening criteria will be scheduled for a second randomization visit. During this visit baseline assessments will be obtained. Eligible subjects will then be randomized to a treatment group and will be provided with the first week's study medications. The goal is to directly compare the efficacy and tolerability of two novel anticonvulsants, zonisamide and levetiracetam, with placebo, and using topiramate, which has extensive evidence supporting its efficacy in alcoholism, as a positive control group. We believe that this will be the first direct comparison of these agents in alcoholism, and the results will provide information on the efficacy and safety of the medications.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, parallel group design study with 4 treatment groups; levetiracetam, zonisamide, topiramate, and placebo control. This study evaluated the effects of zonisamide (400 mg per day) on alcohol consumption and its neurotoxic effects in subjects with AUDS. A double-blind placebo-controlled clinical trial was conducted using two comparator anticonvulsant drugs, topiramate (300 mg daily) and levetiracetam (2000 mg/day), which does not impair cognition. Topiramate was used as an active control in this study.

Study medications were administered for 14 weeks, including a 2-week taper period. Target maintenance doses of study medications were administered to subjects during study weeks 8-12. Dosage reductions were made if needed to allow subjects to tolerate their study medication. During the medication taper phase of the study (Weeks 13-14) the Principal Investigator is allowed flexibility in the titration schedule in instances when the subject is experiencing events consistent with withdrawal, for example anxiety. Neurotoxicity of study drugs was assessed using neuropsychological tests and the AB-Neurotoxicity scale.

An adaptive randomization procedures with sex and heavy drinking history being factors in the assignment of subjects to the treatment groups. will be done using sex and very heavy drinking. Very heavy drinking is defined as male subjects consuming more then 10 standard drinks per day and female subjects consuming more then 8 standard drinks per day for more then 40 percent of the days in the screening TLFB.

Medication adherence was facilitated using Brief Behavioral Compliance Enhancement Treatment. It is a brief, standardized therapy that emphasizes medication adherence as being crucial to the improvement of drinking behavior.

Subject assessments included, but were not limited to the following:

1) TLFB, 2) Adverse Events (AEs) assessment ,3) A-B Neurotoxicity Scale (weeks 1,4,8,12,15),and 4) Neuropsychological battery Assessments- including the Controlled Word Association Test (COWAT) and Digit and Spatial Span portions of the Wechsler Memory Scale- 3rd (weeks 1,12).

ELIGIBILITY:
Inclusion Criteria:

To be admitted into this study candidates must meet the following criteria:

1. DSM-IV-TR Diagnosis of Alcohol Dependence.
2. A minimal level of an average of 28 standard drinks per week for women or 35 drinks per week for men over a baseline 28 day consecutive period prior to the screening session during the 90 day time line follow-back.
3. Male or Female 21- 65 years of age.
4. Able to provide informed consent and comprehend study procedures.
5. Negative urine toxicological screen for opioids, cocaine, amphetamines, methamphetamine, and benzodiazepines. The test may be repeated for opioids or benzodiazepines shown to be medically prescribed for an acute disorder. The urine test may also be repeated if the Investigator deems necessary.
6. A score of >8 on the Alcohol Use Disorder Identification Test (AUDIT) during screening.
7. Must be suitable for outpatient management of alcoholism.
8. Express desire to stop drinking or reduce alcohol consumption.
9. Provide contact information for themselves or an alternate contact that the staff will call in case of missed appointment.
10. Women must be postmenopausal for at least one year, be surgically sterile, or be using an effective method of birth control.
11. Must be able to take oral medications, adhere to the regimen and be willing to return for follow up visits.

Exclusion Criteria:

Subjects meeting the following criteria will be excluded from the study:

1. Dependent on DSM IV-TR drugs or substances other than ethanol, nicotine, or caffeine.
2. DSM IV-TR diagnosis of any current Axis I diagnosis other than alcohol dependence, nicotine dependence, or caffeine dependence that in the opinion of the study physicians might require intervention with either pharmacological or non-pharmacological therapy that will interfere with the course of the study.
3. Receiving inpatient treatment for alcohol dependence, other then alcohol detoxification, within 4 weeks prior to enrollment into this study.
4. Subjects with a score of 10 or greater on the Clinical Institute Withdrawal Assessment for Alcohol-Revised on first or second visits.
5. Being treated with acamprosate, disulfiram or naltrexone within two weeks prior to randomization:
6. Currently being treated with any of the following medications: a) antipsychotic agents. b) antimanic or anticonvulsant agents. c) sedative- hypnotics. d) chronic opioid treatment. e) psychomotor stimulants- amphetamine derivatives, methylphenidate
7. Subjects who are legally mandated to participate in an alcohol treatment program.
8. Use of any medication known to inhibit or induce cytochrome P450 3A4 enzymes.
9. Subjects who have attempted suicide or who have had suicidal ideation within 30 days of their first visit.
10. Subjects with renal disease or history of kidney stones.
11. Subjects with AST or ALT >3 times the upper limit of the normal range during screening.
12. History of significant neurological disorder.
13. Subjects who are pregnant (as assessed by serum HCG) or lactating.
14. Subjects known to have clinically significant medical conditions that in the opinion of the study physician would preclude administration of the study medications or limit participation in the clinical trial.
15. Subjects with history of treatment with levetiracetam, topiramate or zonisamide.
16. Score of 25 or less on the Folstein Mini- Mental examination.
17. History of anticonvulsant-induced rash.
18. Taking drugs that contain "sulfa" moiety, such as sulfonamides, sulfonylureas, carbonic anhydrase inhibitors, thiazides, and loop diuretics (except ethacrynic acid).
19. During the 2 weeks prior to screening subjects who report average drinks per day that are within the guidelines for safe levels of alcohol consumption (i.e. 2 drinks/ day males; 1 drink/day females-HHS standard) will be excluded.
20. Subjects with a sulfa allergy.

    -

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenic A Ciraulo, MD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Knapp CM, Ciraulo DA, Sarid-Segal O, Richardson MA, Devine E, Streeter CC, Oscar-Berman M, Surprise C, Colaneri L, Putnam M, Waters M, Richambault C. Zonisamide, topiramate, and levetiracetam: efficacy and neuropsychological effects in alcohol use disorders. J Clin Psychopharmacol. 2015 Feb;35(1):34-42. doi: 10.1097/JCP.0000000000000246. PMID 25427171

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: Placebo: Matched placebo will be administered orally twice daily beginning on Day 1, Week 1 and continue through Day 7, Week 14.
Period: Overall Study
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Started | 19 | 21 | 21 | 24
Completed | 15 | 17 | 15 | 19
Not Completed | 4 | 4 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill | Total
Number analyzed (Participants) | 19 | 21 | 21 | 24 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 21 | 24 | 85
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (10.0) | 47.5 (10.5) | 46.8 (10.5) | 46.8 (7.3) | 47.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 9 | 11 | 37
  Male | 11 | 12 | 12 | 13 | 48
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 21 | 24 | 85
Education [Mean (Standard Deviation); unit: years] | 15.6 (2.5) | 15.2 (2.4) | 15.4 (1.9) | 15.3 (2.7) | 15.4 (2.4)
Alcohol Use Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — The AUDIT assesses the extent to which an individual exhibits patterns of harmful or hazardous alcohol use. Scale scores for this test can range from 0 to 40, with higher scores indicating greater levels of harmful or hazardous alcohol use.
  units on a scale | 22.1 (5.9) | 23.1 (5.2) | 24.6 (5.7) | 23.7 (4.7) | 23.4 (5.4)
Wechsler Abbreviated Scale of Intelligence (WAIS) [Mean (Standard Deviation); unit: scale scores] — The WASI assesses general cognitive functioning. The Vocabulary and Matrix Reasoning subtests were administered to subjects in this study. The Vocabulary subtest is used to evaluate verbal knowledge, verbal expressiveness, and fund of information. The Matrix Reasoning subtest measures nonverbal reasoning and general intellectual ability. Scores range between 55 to 157, with the higher scores indicating greater intelligence. The mean score for this test is set to be 100.
  scale scores | 115.3 (8.9) | 113.3 (11.6) | 113.6 (12.6) | 110.7 (14.0) | 113.1 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Measure is the Mean Number of Drinks Consumed Per Day Over the Period From Treatment Weeks 10 Through 12 When All Study Medications Should be at Their Maximum Steady Levels Based on Their Known Pharmacokinetic Properties.
Description: Mean standard drinks consumed per day for each treatment week, weeks 10 thru 12. Actual mean values obtained are shown. Analyses are based on model generated least squares means for a two -way repeated measures mixed models analysis for data obtained for weeks 1 through 12, with baseline values used as covariates. Week (time) was used as the within subject factor and treatment group was the between group factor.
Time Frame: Weeks 10, 11, 12
Population: Alcohol dependent subjects. Number of participants analyzed are provided for the number of subjects for data that was available for the timeframe for the specific analyses, i.e. Weeks 10,11,12.
Measure: Mean (Standard Error); unit: Standard Drinks per day
Arm/Group | Zonisamide | Sugar Pill | Topiramate | Levetiracetam
Number analyzed (Participants) | 16 | 20 | 16 | 17
Standard Drinks per day
  Week 10 | 3.8 (0.9) | 6.3 (0.9) | 3.2 (0.8) | 4.6 (0.8)
  Week 11 | 3.4 (0.6) | 6.8 (1.2) | 2.7 (0.7) | 4.3 (0.7)
  Week 12 | 2.5 (0.7) | 6.0 (0.9) | 2.5 (0.7) | 4.3 (0.7)
Statistical Analysis 1: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 10 means for mean drinks per day obtained for the placebo and zonisamide groups. Means used for the analysis are least means squares from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.06, ANOVA — p<0.05 considered to be significant; Difference between least squares means = -2.1, Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 11 means for mean drinks per day obtained for the placebo and zonisamide groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.008, ANOVA — p< 0.05 was considered to be significant; Difference between least squares means = -3.0, Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 12 mean for mean drinks per day obtained for the placebo and zonisamide groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis — p< 0.05 was considered to be significant; Difference between least squares means = -2.1, Standard Error of Mean 1.2
Statistical Analysis 4: Comparison: Sugar Pill vs Topiramate; Comparison of Week 10 mean for mean drinks per day obtained for the placebo and topiramate groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates,; Test type: Superiority or Other; p = 0.003, ANOVA — p<0.05 is considered as being significant; Difference between least squares means. = -3.4, Standard Error of Mean 1.1
Statistical Analysis 5: Comparison: Sugar Pill vs Topiramate; Comparison of Week 11 means for mean drinks per day obtained for the placebo and topiramate groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.0002, ANOVA; Difference between least squares means = -4.4, Standard Error of Mean 1.1
Statistical Analysis 6: Comparison: Sugar Pill vs Topiramate; Comparison of Week 12 means for mean drinks per day obtained for the placebo and topiramate groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.0007, ANOVA; Difference between least squares means = -4.1, Standard Error of Mean 1.2
Statistical Analysis 7: Comparison: Sugar Pill vs Levetiracetam; Comparison of Week 10 means for mean drinks per day obtained for the placebo and levetiracetam groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.15, ANOVA — p<0.05 considered to be significant; Difference between least squares means = -1.64, Standard Error of Mean 1.1
Statistical Analysis 8: Comparison: Sugar Pill vs Levetiracetam; Comparison of Week 11 means for mean drinks per day obtained for the placebo and levetiracetam groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariate values; Test type: Superiority or Other; p = 0.014, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -2.9, Standard Error of Mean 1.2
Statistical Analysis 9: Comparison: Sugar Pill vs Levetiracetam; Comparison of Week 12 means for mean drinks per day obtained for the placebo and levetiracetam groups. Means used for the analysis are least squares means s from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.1, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -2.0, Standard Error of Mean 1.2

2. Secondary Outcome: AB-Neurotoxicity Scale.
Description: Total Scores AB-Neurotoxicity Scale Week 12. This scale provides subject ratings of anticonvulsant neurotoxic effects. Scores may range 0 to 72, with possibility of an additional 30 points being for complaints not listed in the list of complaints provides. Total scores, therefore, may be as high as 102, with higher scores indicating greater severity of problems. Actual mean scores are shown. Means for the analysis are least means squares values obtained from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates.
Time Frame: Week 12
Population: Alcohol dependent subjects.
Measure: Mean (Standard Error); unit: Scale Scores
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Number analyzed (Participants) | 15 | 17 | 15 | 19
Scale Scores | 7.1 (2.2) | 11.3 (2.7) | 15.4 (3.3) | 5.8 (1.6)
Statistical Analysis 1: Comparison: Topiramate vs Sugar Pill; Comparison between mean values obtained for the topiramate and placebo groups for Week 12. Model generated least mean squares were used for this analysis; Test type: Superiority or Other; p = 0.015, ANOVA — p< 0.05 is considered to be significant; Mean difference Week 12 = 8.9, Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: Zonisamide vs Sugar Pill; Comparison of means for the zonisamide and placebo group for Week 12. Mixed models generated means were used in this analysis; Test type: Superiority or Other; p = 0.784, ANOVA — p< 0.05 is considered to be significant; Mean Difference Week 12 = 0.98, Standard Error of Mean 3.6
Statistical Analysis 3: Comparison: Levetiracetam vs Sugar Pill; Comparison of means for the levetiracetam and placebo groups for Week 12. Model generated least mean squares were used for this analysis; Test type: Superiority or Other; p = 0.264, ANOVA — p< 0.05 is considered to be significant; Mean difference Week 12 = 3.65, Standard Error of Mean 3.3

3. Secondary Outcome: Mean Percent Days Heavy Drinking
Description: Mean weekly values for each treatment group for percent days heavy drinking. Heavy drinking was defined as 4 or more drinks per day for women and 5 or more drinks per day for men.
Time Frame: Weeks 10, 11, 12
Population: Alcohol dependent subjects. Alcohol dependent subjects. Number of participants analyzed are provided for the number of subjects for data that was available for the time frame for the specific analyses, i.e. Weeks 10,11,12.
Measure: Mean (Standard Error); unit: Percentage of Days/Week
Arm/Group | Zonisamide | Sugar Pill | Topiramate | Levetiracetam
Number analyzed (Participants) | 16 | 20 | 16 | 17
Percentage of Days/Week
  Week 10 | 38.4 (10.7) | 65.7 (6.5) | 32.1 (8.5) | 49.6 (9.4)
  Week 11 | 36.6 (8.5) | 61.7 (8.1) | 29.5 (7.1) | 47.9 (9.3)
  Week 12 | 34.3 (11.0) | 60.9 (8.0) | 21.0 (8.1) | 44.5 (8.7)
Statistical Analysis 1: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 10 means for mean percent heavy drinking days obtained for the placebo and zonisamide groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.013, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -24.4, Standard Error of Mean 9.7
Statistical Analysis 2: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 11 means for mean percent heavy drinking days obtained for the placebo and zonisamide groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.036, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -20.9, Standard Error of Mean 9.8
Statistical Analysis 3: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 12 means for mean percent heavy drinking days obtained for the placebo and zonisamide groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.24, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -22.8, Standard Error of Mean 9.9
Statistical Analysis 4: Comparison: Sugar Pill vs Topiramate; Comparison of Week 10 means for mean percent heavy drinking days obtained for the placebo and topiramate groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.0004, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -33.0, Standard Error of Mean 9.0
Statistical Analysis 5: Comparison: Sugar Pill vs Topiramate; Comparison of Week 11 means for mean percent heavy drinking days obtained for the placebo and topiramate groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.0015, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -29.7, Standard Error of Mean 9.2
Statistical Analysis 6: Comparison: Sugar Pill vs Topiramate; Comparison of Week 12 means for mean percent heavy drinking days obtained for the placebo and topiramate groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p < 0.0001, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -37.7, Standard Error of Mean 9.3
Statistical Analysis 7: Comparison: Sugar Pill vs Levetiracetam; Comparison of Week 10 means for mean percent heavy drinking days obtained for the placebo and levetiracetam groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.04, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -20.7, Standard Error of Mean 10.0
Statistical Analysis 8: Comparison: Sugar Pill vs Levetiracetam; Comparison of Week 11 means for mean percent heavy drinking days obtained for the placebo and levetiracetam groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.025, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -23.3, Standard Error of Mean 10.2
Statistical Analysis 9: Comparison: Sugar Pill vs Levetiracetam; Comparison of Week 12 means for mean percent heavy drinking days obtained for the placebo and levetiracetam groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.018, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -24.8, Standard Error of Mean 10.3

4. Secondary Outcome: Percent Days Drinking
Description: Mean percent days drinking for Weeks 10, 11, 12. A drinking day is considered to be a day in which 1 or more drinks have been consumed. Means are model generated least means squares values obtained from a two-way repeated measures analysis from data obtained from Weeks 1 through 12, with Week as the within subject factor and treatment group as the between group factor.
Time Frame: Weeks 10, 11, 12
Population: Alcohol dependent subjects. Alcohol dependent subjects. Number of participants analyzed are provided for the number of subjects for data that was available for the timeframe for the specific analyses, i.e. Weeks 10,11,12.
Measure: Mean (Standard Error); unit: Percentage of Days/ Week
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Number analyzed (Participants) | 15 | 17 | 15 | 19
Percentage of Days/ Week
  Week 10 | 61.6 (9.5) | 72.2 (8.3) | 51.8 (10.1) | 83.6 (5.2)
  Week 11 | 62.1 (9.3) | 68.9 (8.6) | 43.8 (9.6) | 87.2 (5.1)
  Week 12 | 61.3 (9.9) | 73.1 (7.6) | 51.4 (11.0) | 78.2 (6.2)
Statistical Analysis 1: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 10 means for mean percent drinking days obtained for the placebo and zonisamide groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.005, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -22.5, Standard Error of Mean 7.8
Statistical Analysis 2: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 11 means for mean percent drinking days obtained for the placebo and zonisamide groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.003, ANOVA; Difference between least squares means = -24.1, Standard Error of Mean 7.9
Statistical Analysis 3: Comparison: Zonisamide vs Sugar Pill; Comparison of Week 12 means for mean percent drinking days obtained for the placebo and zonisamide groups Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.044, ANOVA — p< 0.05 is considered to be significant; Difference between least square means = -16.3, Standard Error of Mean 8.0
Statistical Analysis 4: Comparison: Topiramate vs Sugar Pill; Comparison of Week 10 means for mean percent drinking days obtained for the placebo and topiramate. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factors. Baseline values were used as covariates; Test type: Superiority or Other; p < 0.0001, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -38.1, Standard Error of Mean 9.0
Statistical Analysis 5: Comparison: Topiramate vs Sugar Pill; Comparison of Week 11 means for mean percent drinking days obtained for the placebo and topiramate. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p < 0.0001, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -47.6, Standard Error of Mean 9.1
Statistical Analysis 6: Comparison: Topiramate vs Sugar Pill; Week 12.Comparison of Week 12 means for mean percent drinking days obtained for the placebo and topiramate. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis, with Week (time) as the the within subject factor and treatment as the between group factor. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.0004, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -34.0, Standard Error of Mean 9.2
Statistical Analysis 7: Comparison: Levetiracetam vs Sugar Pill; Comparison of Week 10 means for mean percent drinking days obtained for the placebo and levetiracetam groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.017, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -19.3, Standard Deviation 8.0
Statistical Analysis 8: Comparison: Levetiracetam vs Sugar Pill; Comparison of Week 11 means for mean percent drinking days obtained for the placebo and levetiracetam groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis. Baseline values were used as covariates; Test type: Superiority or Other; p = 0.0002, ANOVA — p<0.05 is considered to be significant; Difference between least squares means = -31.2, Standard Error of Mean 8.1
Statistical Analysis 9: Comparison: Levetiracetam vs Sugar Pill; .Comparison of Week 12 means for mean percent drinking days obtained for the placebo and levetiracetam groups. Means used for the analysis are least squares means from a two-way repeated measures mixed models analysis.Baseline values were used as covariates; Test type: Superiority or Other; p = 0.026, ANOVA — p< 0.05 is considered to be significant; Difference between least squares means = -18.5, Standard Error of Mean 8.2

5. Secondary Outcome: Controlled Word Association Test (COWAT)- Letter Fluency
Description: Number of words generated that start with a set of 3 letters. The COWAT provides a measure of verbal fluency. Actual means for COWAT results are shown.
Time Frame: Baseline & Week 12
Population: Alcohol Dependent Subjects. Number of participants analyzed represent the number for whom Week 12 data was available.
Measure: Mean (Standard Error); unit: Number of Words Produced
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Number analyzed (Participants) | 13 | 17 | 15 | 17
Number of Words Produced
  Baseline | 46.5 (3.1) | 46.2 (3.0) | 43.4 (3.8) | 47.4 (2.8)
  Week 12 | 32.5 (2.2) | 45.4 (2.7) | 28.1 (2.0) | 50.5 (2.4)
Statistical Analysis 1: Comparison: Zonisamide vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that COWAT-Letter Fluency scores would change towards a downward direction for the zonisamide as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p< 0.01 is considered to be significant; p value is for the group x time interaction term.'
Statistical Analysis 2: Comparison: Topiramate vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that COWAT-Letter Fluency scores would change towards a downward direction for the topiramate as compared to the placebo group resulting in a significant treatment x time interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p<0.01 is considered to be significant; p value is for group x time interaction term for the comparison of data for the topiramate and placebo group
Statistical Analysis 3: Comparison: Levetiracetam vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that COWAT-Letter Fluency scores would change towards a downward direction for the levetiracetam as compared to the placebo group resulting in a significant treatment x time interaction; Test type: Superiority or Other; p = 0.30, Mixed Models Analysis — p<0.01 is considered to be significant; p value is for interaction effect for the comparison of data for the levetiracetam and placebo groups

6. Secondary Outcome: COWAT-Category
Description: Number of words produced by subjects over 60 seconds for a semantic category (Animals). The COAWAT-Category sub-test provides a measure of verbal fluency. Mean value shown are actual means for the number of words produced.
Time Frame: Baseline, Week12
Population: Alcohol Dependent Subjects. Number of participants analyzed represent the number for whom Week 12 data was available.
Measure: Mean (Standard Error); unit: Number of Words Produced
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Number analyzed (Participants) | 13 | 17 | 15 | 17
Number of Words Produced
  Baseline | 22.6 (1.1) | 20.9 (0.9) | 21.9 (1.3) | 21.6 (1.2)
  Week 12 | 17.4 (0.7) | 21.2 (1.0) | 17.0 (1.2) | 20.8 (0.7)
Statistical Analysis 1: Comparison: Zonisamide vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that COWAT-Category scores would change towards a downward direction for the zonisamide as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — p<0.01 is considered to be significant; p value is for the group x time interaction effect for the paired comparison of COWAT-category data for the zonisamide and placebo groups
Statistical Analysis 2: Comparison: Topiramate vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that COWAT-Category scores would change towards a downward direction for the topiramate as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — p< 0.01 is considered to be significant; The p value shown is for the group x time interaction effect for the comparison of data from the topiramate and the placebo groups
Statistical Analysis 3: Comparison: Levetiracetam vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that COWAT-Category scores would change towards a downward direction for the levetiracetam as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p = 0.36, Mixed Models Analysis — p<0.01 is considered to be significant; The p value is for the group x time interaction effect for the comparison of the levetiracetam and placebo groups

7. Secondary Outcome: Wechsler Memory Scales (WMS)-3d Ed Digit Span-Age Adjusted Total
Description: WMS Digit Span is a measure of working memory. Subjects respond by repeating lists of number sequences presented by the test administrator. Age adjusted scores are presented below. Scores may range between 1 and 19, with lower scores indicating poorer performance on the task.
Time Frame: Baseline, Week 12
Population: Alcohol Dependent Subjects. Number of participants analyzed represent the number for whom Week 12 data was available.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Number analyzed (Participants) | 13 | 17 | 15 | 17
units on a scale
  Baseline | 11.8 (0.8) | 11.9 (0.7) | 12.1 (0.6) | 12.6 (0.7)
  Week 12 | 10.0 (0.9) | 12.2 (0.8) | 7.7 (0.6) | 13.0 (0.9)
Statistical Analysis 1: Comparison: Zonisamide; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that Digit span scores would change towards a downward direction for the zonisamide as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis — p<0.01 is considered to be significant; p value is for the group x time interaction effect
Statistical Analysis 2: Comparison: Topiramate vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that age adjusted Digit Span scores would change towards a downward direction for the topiramate as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p<0.01 is considered to be significant; p value shown is for the group X time interaction effect
Statistical Analysis 3: Comparison: Levetiracetam vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that Digit span scores would change towards a downward direction for the levetiracetam as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p = 0.95, Mixed Models Analysis — p<0.01 is considered to be significant; p value shown is for the group x time interaction effect

8. Secondary Outcome: Wechsler Memory Scale-3rd Ed. Spatial Span
Description: WMS Spatial Span test measures working memory for a spatial sequence of numbers. This assesses visual working memory. Age adjusted scaled scores are presented. Score may range between 1 and 19, with lower scores indicating greater impairment in performance.
Time Frame: Baseline, Week 12
Population: Alcohol Dependent Subjects. Number of participants analyzed represent the number for whom Week 12 data was available.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Number analyzed (Participants) | 13 | 17 | 15 | 17
units on a scale
  Baseline | 10.8 (0.7) | 10.5 (0.6) | 12.0 (0.6) | 10.8 (0.8)
  Week 12 | 7.9 (0.9) | 10.9 (0.5) | 8.4 (0.7) | 10.4 (0.8)
Statistical Analysis 1: Comparison: Zonisamide vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that Spatial Span scores would change towards a downward direction for the zonisamide as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis — p<0.01 is considered to be significant; p value shown is for the group x time effect
Statistical Analysis 2: Comparison: Topiramate vs Sugar Pill; Data were analyzed using two-way repeated measures mixed models analysis. It was hypothesized that Digit span scores would change towards a downward direction for the topiramate as compared to the placebo group resulting in significant treatment x time interaction; Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis — p<0.01 is considered to be significant; p value shown is for the group x time interaction effect
Statistical Analysis 3: Comparison: Levetiracetam vs Sugar Pill; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis — p<0.01 is considered to be significant; p value shown is for the group x time interaction effect

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of 17 weeks for each subject and for a total of throughout the entire study.
Arm/Group | Zonisamide | Levetiracetam | Topiramate | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/21 | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 15/19 | 11/21 | 13/21 | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=19) | Levetiracetam (N=21) | Topiramate (N=21) | Sugar Pill (N=24)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 | 0 | 0 — Rated as being only remotely to zonisamide use.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=19) | Levetiracetam (N=21) | Topiramate (N=21) | Sugar Pill (N=24)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Altered Taste (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased Libido (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Dissociation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disoriented (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erectile Dsyfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fatigue (Nervous system disorders) | 3 (3) | 5 (5) | 2 (2) | 3 (3)
GI Distress (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 6 (6) | 4 (4) | 2 (2)
Impaired Concentration (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Impaired Memory (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Irritability (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Lightheaded (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of Appetite (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Prurtitus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Slowed Thinking (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight Loss (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Word Finding (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination lead to a small number of subjects in each group being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No